CLINICAL TRIAL: NCT05047406
Title: Effect of Probiotic Administration on Infection Incidence Rate in Living Donor Liver Transplantation Recipients
Brief Title: Bacillus Clausii in Liver Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Ezzeldin Nabet, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RHDIRB2020110301REC 46
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Transplantation Infection; Liver Grafting; Hepatic Transplantation
Keywords: liver; transplantation; infection; probiotics; Bacillus clausii
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, open-label, parallel, single-center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): 2 oral mini-bottles daily of Bacillus clausii probiotic liquid containing 2 billion spores/bottle for 2 weeks before living donor liver transplantation surgery In addition, patients will receive standard of care regarding immunosuppressants and antibiotic prophylaxis
  Interventions: Dietary Supplement: Bacillus clausii Probiotic liquid
- Control (No Probiotic) (No Intervention): patients will receive standard of care regarding immunosuppressants and antibiotic prophylaxis

INTERVENTIONS:
Dietary Supplement: Bacillus clausii Probiotic liquid — mini bottles for oral administration containing 2 million spores of Bacillus clausii
  Other Names: Enterogermina
  Arms: Probiotic

SUMMARY:
A prospective, randomized, controlled study of the safety and efficacy of using Bacillus clausii probiotic oral preparation to decrease the incidence of infection during the first 30 days after living donor liver transplantation surgery.

DETAILED DESCRIPTION:
Patients planned for living donor liver transplantation would be randomized to either intervention or control group 2 weeks before surgery. Intervention group shall receive Bacillus clausii probiotics for 2 weeks. patients in both groups would be followed-up for adverse events and signs and symptoms of infection up to 30 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 - 65 years.
* Patients suffering from end stage liver disease (ESLD) with any etiology listed on waiting list and accepting to volunteer in the study with the informed consent.
* Patients not suffering from any active infection at the start of the study.

Exclusion Criteria:

* Patients with poorly controlled autoimmune disease on immunosuppression before transplantation.
* Patients who undergo combined kidney-liver transplantation.
* Patients with severe renal insufficiency (creatinine clearance <50 ml/min).
* Patients with intestinal obstruction (ileus).
* Patients with cerebral disorders with danger of aspiration.
* Patients with roux en Y-anastomosis.
* Patients with cystic fibrosis.
* Retransplantation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
infection and mortality rates | up to 30 days post-operatively
  the occurrence of post-operative bacterial infection and mortality

SECONDARY OUTCOMES:
type of isolated bacteria | up to 30 days post-operatively
  culture and sensitivity results of isolated bacteria
total hospital stay | up to 30 days post-operatively
  total length of hospital stay defined as the day of surgery and day of discharge
total ICU stay | up to 30 days post-operatively
  total length of ICU stay defined as the day of surgery and day of regular ward transfer
Incidence of Probiotic related adverse events | starting 2 weeks before surgery and up to 30 days post-operatively
  incidence of adverse events and/or side effects related to probiotics use
Duration of antibiotic therapy | up to 30 days post-operatively
  duration of antibiotic therapy after exclusion of period of antibiotic prophylaxis without signs of infection
quality of life assessment | at baseline, on day 15 before surgery, and at 30 days post-transplantation
  quality of life assessment using liver disease symptom index 2.0 questionnaire
Aspartate aminotransferase level (AST) | at baseline before probiotic administration and at 30 days post-transplantation
  serum aspartate aminotransferase level
Alanine aminotransferase level (ALT) | at baseline before probiotic administration and at 30 days post-transplantation
  serum alanine aminotransferase level
international normalized ratio | at baseline before probiotic administration and at 30 days post-transplantation
  ratio between patient's prothrombin time and that of health laboratory standard
Total bilirubin level | at baseline before probiotic administration and at 30 days post-transplantation
  total serum bilirubin level

CONTACTS AND LOCATIONS:
Overall Officials: Rana Sayed, PhD, Study Director — Faculty of Pharmacy, Ain Shams University
Locations (1):
- Ain Shams Center for Organ Transplantation, Ain Shams Specialized Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No